CLINICAL TRIAL: NCT03598452
Title: A Prospective, Non-randomized, Non-controlled Trial: Initial Intravitreal Injection of High-dose Ganciclovir for Cytomegalovirus Retinitis in HIV-negative Patients
Brief Title: High-dose Intravitreal Injection of Ganciclovir for the Treatment of CMVR in HIV-negative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHIRB2018017
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Infection Viral; Uveitis, Posterior
Keywords: Cytomegalovirus retinopathy; High-dose; Ganciclovir; Intravitreal injection
MeSH Terms: conditions — Virus Diseases; Uveitis, Posterior; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High dose of ganciclovir group (Experimental): IVG was conducted in a week interval. The initial dose was 6mg/0.1ml at the first injection and it was reduced to 4.5mg/0.1ml at the second time; 3mg/0.1ml of IVG was maintained until the CMV could not be detected in aqueous humor.
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir — Intravitreal Injection of Ganciclovir (IVG) was conducted in a week interval. The initial dose was 6mg/0.1ml at the first injection and it was reduced to 4.5mg/0.1ml at the second time; 3mg/0.1ml of IVG was maintained until the CMV could not be detected in aqueous humor.

SUMMARY:
This prospective, non-randomized, non-controlled clinical trial was conducted to examine the clinical outcomes achieved by using initial high-dose intravitreal ganciclovir injections of ganciclovir in treating cytomegalovirus (CMV) retinitis in patients without human immunodeficiency virus (HIV) infection.

DETAILED DESCRIPTION:
Cytomegalovirus retinitis (CMVR) is a serious vision-threatening disease. Intravitreal antiviral drug delivery was used as first-line treatment in several studies when systematic injection has been ruled out. The reported dose of intravitreal injections of ganciclovir (IVG) varied from 200 μg/0.1 ml to 5mg/0.1 ml in patients with AIDS. There was no consensus on the dose of ganciclovir in the treatment of CMVR in HIV-negative patients. Previous work showed the safety and the efficacy of 1mg IVG. The investigators proposed that a higher dose of ganciclovir (6mg/0.1ml) for the first injection followed by lower dose for maintenance may indicate a better result. Therefore, this study was performed to evaluate the therapeutic effect and safety of initial high-dose IVG for CMVR in HIV-negative patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CMVR by ophthalmological examination
* Positive CMV-DNA in aqueous humor approved by real-time PCR.
* HIV-negative.

Exclusion Criteria:

* Diabetic retinopathy,
* Glaucoma.
* Optic neuritis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
CMV-DNA load in aqueous humor | Once a week. From the date of the first IVG until the date in which the CMV-DNA load turned undectable, assessed up to 10 weeks.
  The load of CMV-DNA level in aqueous humor was detected by means of real-time polymerase chain reaction (PCR). The aqueous humor was obtained before the IVG.

SECONDARY OUTCOMES:
Visual function | Once a week. From the date of the first IVG until the date in which the CMV-DNA load turned undectable, assessed up to 10 weeks.
  Best corrected visual acuity (BCVA) measured using a decimal chart
Occurrence of IVG-related complications | Once a week. From the date of the first IVG until the date in which the CMV-DNA load turned undectable, assessed up to 10 weeks.
  The occurence of IVG-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Doctor, Study Director — Shanghai Aier Eye Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The accurate CMV-DNA load and its change will be shared in the published paper.

REFERENCES:
- [Background] Jeon S, Lee WK, Lee Y, Lee DG, Lee JW. Risk factors for cytomegalovirus retinitis in patients with cytomegalovirus viremia after hematopoietic stem cell transplantation. Ophthalmology. 2012 Sep;119(9):1892-8. doi: 10.1016/j.ophtha.2012.03.032. Epub 2012 May 30. PMID 22657564
- [Background] Kuo IC, Kempen JH, Dunn JP, Vogelsang G, Jabs DA. Clinical characteristics and outcomes of cytomegalovirus retinitis in persons without human immunodeficiency virus infection. Am J Ophthalmol. 2004 Sep;138(3):338-46. doi: 10.1016/j.ajo.2004.04.015. PMID 15364214
- [Result] Miao H, Tao Y, Jiang YR, Li XX. Multiple intravitreal injections of ganciclovir for cytomegalovirus retinitis after stem-cell transplantation. Graefes Arch Clin Exp Ophthalmol. 2013 Jul;251(7):1829-33. doi: 10.1007/s00417-013-2368-6. Epub 2013 May 12. PMID 23665863
- [Derived] Qian Z, Li H, Tao Y, Li W. Initial intravitreal injection of high-dose ganciclovir for cytomegalovirus retinitis in HIV-negative patients. BMC Ophthalmol. 2018 Dec 10;18(1):314. doi: 10.1186/s12886-018-0983-z. PMID 30526535